CLINICAL TRIAL: NCT01431248
Title: Preterm Premature Rupture of Membranes: Erythromycin Versus Azithromycin. A Randomized Trial Comparing Their Efficacy to Prolong Latency
Brief Title: PPROM Erythromycin Versus Azithromycin
Acronym: PEACE
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: PEACE
Record Dates: First submitted 2011-09-07; First posted 2011-09-09 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Preterm Premature Rupture of Membranes
Keywords: Preterm Premature Rupture of Membranes; Erythromycin; Azithromycin
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Azithromycin: Azithromycin 1gm PO once
- Erythromycin 250mg: Erythromycin 250mg IV Q 6hrs x 48 hours followed by 500 mg PO Q 8 hours x 5 days.

SUMMARY:
Preterm Premature Rupture of Membranes (PPROM) is treated with an antibiotic, erythromycin or azithromycin, to prolong pregnancy. Erythromycin is taken for several days and can result in stomach upset in some patients, causing them to stop taking the medication. Therefore, azithromycin is often prescribed instead. Azithromycin is usually taken only once and stomach upset is not seen or greatly reduced. The goal of this study is to see if there is a difference between the antibiotic (azithromycin) compared to the antibiotic (erythromycin) in prolonging pregnancy in patients with Preterm Premature Rupture of Membranes (PPROM). The working hypothesis is that there is no difference in the clinical effectiveness between antibiotic regimens containing te macrolides azithromycin and erythromycin for prolonging latency in PPROM.

DETAILED DESCRIPTION:
The current standard regimen for PPROM patients between the gestational age of 24 0/7 and 32 0/7 weeks, is to administer ampicillin 2gm IV every 6hours for 48hrs followed by amoxicillin 250mg orally every 8 hours for 5 days, with erythromycin 250mg IV for 48hours followed by 500mg orally every 8hours for 5 days. Our study design would be a prospective randomized trial. Consented, eligible women will be randomized to receive ampicillin as above plus either azithromycin 1 gm orally at enrollment or erythromycin 250mg IV every 6 hours for 48hours followed by 500mg orally every 8hours for 5 days. Those who are unable to tolerate the 1gm of azithromycin within the first 30 minutes of administration, a 1000mg powder suspension will be given. In conjunction with standard protocol, a course of steroids for fetal lung maturity will be administered upon the treating staff's discretion, and all Group B Beta Streptococcus positive patients will be treated.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at least 18 years old
* Gestational age of 24 0/7 to 32 0/7 weeks
* Singleton gestation
* Randomization within 36 hours of rupture of membranes.
* Cervical dilation less than or equal to 4 cm.

Exclusion Criteria:

* Known lethal fetal anomaly
* Vaginal bleeding
* Maternal or fetal indication for delivery
* Diagnosis of chorioamnionitis on admission
* Cervical cerclage in place
* Placenta previa or other known placental anomalies
* Use of antibiotic therapy within 5 days.
* Allergy or other contraindications to erythromycin/azithromycin or steroid use.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with the diagnosis of PPROM will be enrolled in this protocol.
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Time to delivery | 2 years
  To compare the mean time to delivery, using azithromycin versus erythromycin to prolong latency in PPROM patients. The working hypothesis for this aim is that there is no difference in the clinical effectiveness between antibiotic regimens containing the macrolides azithromycin and erythromycin for prolonging latency in PPROM.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Knudtson, MD, Principal Investigator — University of Oklahoma